CLINICAL TRIAL: NCT04307446
Title: The Feasibility of Immersive Virtual Reality as a Treatment for Chronic Back Pain
Brief Title: Immersive Virtual Reality and Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Nancy Baker, Associate Professor, Tufts University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000192; UL1TR002544 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 10 Minutes/20 Minutes (Experimental): Subject takes part in 10 minute VR experience first and 20 minute VR experience second
  Interventions: Device: Immersive Virtual Reality
- 20 Minutes/10 Minutes (Experimental): Subject takes part in 20 minute VR experience first and 10 minute VR experience second
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Immersive Virtual Reality

SUMMARY:
In the proposed project the investigators will evaluate the feasibility of Immersive Virtual Reality (IVR) and assess the initial effects of IVR on symptoms, affect, and tolerance to cutaneous stimuli. In this single-arm trial, the investigators will recruit 20 adults with CBP. Prior to their IVR experience, subjects will complete multiday baseline assessments using ecological momentary assessment (EMA) methodology to establish typical levels of symptoms and affect. Afterward, in a single experimental session, they will participate in two counterbalanced IVR sessions: one 10-minute and one 20-minute. Immediately after each session the investigators will measure current symptoms and affect using valid and reliable self-report questionnaires, and we will measure changes in tolerance to cutaneous stimuli using quantitative sensory testing. We will measure symptoms and affect for 72 hours after the experimental session using EMA to determine if there is a carryover. At the completion of this study, we will continue to work with stakeholders to develop clinically relevant IVR interventions for people with CBP.

DETAILED DESCRIPTION:
Visit 1-Remote: Consent. Random assignment: Subjects will complete informed consent and data collection of baseline information (demographics, medical history, perceptions of pain, and experiences with VR), surveys on pain, Pain interference, fatigue, and affect. The investigators will also help the participant upload the EMA technology onto their personal phone or tablet. Subjects will then be randomly assigned to receive either the 10- minute IVR session first or the 20-minute IVR session first. Visit 1 will take between 45 and 60 minutes.

Multiple Baseline EMA-Remote: Visit 2 will be scheduled 1-2 weeks later. During the time between visits the investigators will use ecological momentary assessment (EMA) technology to collect multiple measures of pain, fatigue and affect. In EMA subjects respond to prompts delivered through their cell phone or tablet ("pings") with documentation of current symptoms. It is a well-recognized method to capture immediate, synchronized experiences in subjects' natural environments. During this data collection period subjects will be "pinged" 3x daily and asked to rate their current levels of pain, fatigue, and affect. Time to complete these responses will be 15 minutes.

Visit 2-In person: pre Survey/Quantitative Sensory Testing (QST); First VR visit; post Survey/QST. The investigators will collect current pain, pain interference, fatigue and affect, and Quantitative Sensory Testing (QST). QST involves cutaneous (skin) psychophysical (semi-subjective) testing to assess sensory and pain perception pathways. QST quantifies the thresholds of detection of stimuli, the perceived intensity, and the temporal summation (changes in perception over multiple applications). These pain testing procedures are widely-accepted, non-invasive, and non-tissue damaging. The investigators will complete two types QST. Mechanical Pressure Pain Thresholds (MPPTh) will be assessed using a digital pressure algometer on the right upper trapezius and right thumb MP joint. Mechanical Temporal Summation of Pain (MTSP) will be assessed using weighted pinprick stimulators. The investigators will apply a train of 10 stimuli at the rate of 1 per second on the middle finger of the right hand, and subjects will rate the painfulness of the first, fifth, and tenth stimulus. All subjects will take part in two VR experiences (10 min and 20 min) for a total of 30-minutes in VR. After each experience subjects will rate their current pain, fatigue, and affect, and the investigators will complete QST. At the end of both sessions the subjects will rate their experiences of immersion using the Igroup Presence Questionaire, engagement using the Use Engagement Scale (UES), and simulation tolerance using the Simulator Sickness Questionnaire (SSQ). The investigators will also ask a series of open-ended questions about the participant's experiences with IVR and participation in the study. These will include questions about their enjoyment, perceptions of pain, and what they liked/did not like about the IVR experience as well as questions about the burden of being in the study. Visit 2 will take 1.5 to 2 hours

Post Visit 2 EMA-Remote: Subjects will complete three more days (72 hours) of 3x a day prompts for pain, fatigue and affect.

Visit 3-In person: pre Survey/Quantitative Sensory Testing (QST); Second VR visit; post Survey/QST

Post Visit 3 EMA-Remote: Subjects will complete 2 more days (48 hours) of 3x a day prompts for pain, fatigue and affect.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 75 years old
2. Any Back Pain (including neck pain) that has lasted greater than 3 months due to non-cancer related injury or illness.

Exclusion Criteria:

1. People with back pain primarily due to rheumatic (e.g. rheumatoid arthritis or fibromyalgia)
2. people with back pain due to central neurological disorders (e.g. stroke, multiple sclerosis, spinal cord injury)
3. has contagious disorder on the face (such as pink eye) that could be transmitted via the VR head set or has open areas on the face that would come in contact with the headset
4. had a seizure, loss of awareness, or other symptom linked to an epileptic condition
5. insufficient vision to see IVR programs
6. insufficient upper extremity coordination to operate IVR controls
7. insufficient cognitive ability to answer questionnaires or learn to use the IVR
8. unable to understand and respond to English
9. Does not own a cell phone or tablet for baseline and follow-up EMA testing.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Baker, ScD, Principal Investigator — Tufts University
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 Minutes/20minutes: Subject takes part in 10 minute VR experience first and a 20 minute VR experience second
  Immersive Virtual Reality: Immersive Virtual Reality
- 20 Minutes/10 Minutes: Subject takes part in 20 minute VR experience first and a 10 minute VR experience second
  Immersive Virtual Reality: Immersive Virtual Reality
Period: Overall Study
Arm/Group | 10 Minutes/20minutes | 20 Minutes/10 Minutes
Started | 12 | 11
Completed | 10 | 11
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Minutes/20minutes | 20 Minutes/10 Minutes | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (18.6) | 44.8 (14.5) | 49.7 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 9 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
Length of Pain [Mean (Standard Deviation); unit: years] | 12.8 (14.1) | 14.9 (15.8) | 13.9 (15.0)
Previous IVR Experience [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 7 | 6 | 13
  Don't Know | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Numerical Rating Scale
Description: Pain Intensity - Numerical rating scale 0 to 10 with lower score better score
Time Frame: Change in Pain Intensity from before to immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 10 Minutes VR: Received 10 minutes of VR (regardless of order)
- 20 Minutes: 20 minutes of VR regardless of order
Arm/Group | 10 Minutes VR | 20 Minutes
Number analyzed (Participants) | 21 | 20
units on a scale | 0.8 (3.1) | 1.1 (2.2)

2. Primary Outcome: Mechanical Pressure Pain Thresholds (MPPTh)
Description: Sensitivity to pressure will be assessed using a digital pressure algometer on the right upper trapezius and right thumb MP joint. The measures from each site were averaged to obtain an overall mean pressure score for each participant. A lower score indicates a better outcome.
Time Frame: Median Pre and post intervention sensitivity to pressure scores in kilograms
Measure: Median (Full Range); unit: kilograms
Arm/Group | 10 Minutes VR | 20 Minutes
Number analyzed (Participants) | 21 | 20
kilograms
  Pre Intervention | 5.0 [2.5 to 9.6] | 5.0 [2.5 to 8.8]
  Post Intervention | 4.9 [2.6 to 8.4] | 5.1 [3.1 to 8.2]

3. Primary Outcome: Mechanical Temporal Summation of Pain (MTSP)
Description: Sensitivity to pinprick was assessed using weighted pinprick stimulators. We applied a train of 10 stimuli at the rate of 1 per second on the middle finger of the right hand, and subjects rated the painfulness of the first and tenth stimulus using a 1 to 100 pain intentsity rating scale. We calculated the difference from the 1st stimuus to the 10th stimulus to calculate the sensitivity. A lower change score is a better outcome
Time Frame: Change in Sensitivity to pinprick from before to immediately after intervention
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 10 Minutes VR | 20 Minutes
Number analyzed (Participants) | 21 | 20
units on a scale
  Pre Intervention | 8.5 [1 to 40] | 10.0 [-0.5 to 47.5]
  Post Intervention | 8.8 [-2 to 31] | 8.8 [-2.5 to 65]

4. Secondary Outcome: PANAS
Description: Two scales one for Positive and one for Negative Affect - Score for each scale 10 to 50 with lower score indicating less of that affect
Time Frame: Change in affect form before immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 Minutes VR | 20 Minutes
Number analyzed (Participants) | 21 | 20
units on a scale
  PANAS Positive | -1.1 (2.3) | -0.8 (3.3)
  PANAS Negative | -0.7 (2.4) | -0.1 (1.9)

5. Secondary Outcome: PROMIS Fatigue
Description: Fatigue on a scale of 0 to 28 with a lower score indicating less frequent experiences of fatigue
Time Frame: Change in fatigue from before to immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 Minutes VR | 20 Minutes
Number analyzed (Participants) | 21 | 20
units on a scale | 0.1 (1.3) | -0.5 (0.8)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: No difference
Groups:
- 10 Minutes: Subject takes part in 10 minute VR experience regardless of order
  Immersive Virtual Reality: Immersive Virtual Reality
- 20 Minutes: Subject takes part in 20 minute VR experience regardless of order
  Immersive Virtual Reality: Immersive Virtual Reality
Arm/Group | 10 Minutes | 20 Minutes
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04307446/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT04307446/ICF_001.pdf